CLINICAL TRIAL: NCT07290296
Title: Popliteus Muscle Release Versus Kinesio Taping on Patellofemoral Pain Syndrome
Brief Title: Popliteus Muscle Release Versus Kinesio Taping
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hafsa Hesham Abdullah, Physical Therapist, MSc in Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/005805
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): The control group will receive traditional physical therapy treatment at the painful anterior knee, which includes quadriceps strength, hip abduction strength, hip extension strength, hamstring stretch, and gait training.
  Interventions: Other: Traditional Physical Therapy Treatment
- Study Group 1 (Active Comparator): Study group 1 will receive traditional treatment as the control group plus release to the popliteus muscle.
  Interventions: Other: Traditional Physical Therapy Treatment; Other: Popliteus Muscle Release
- Study Group 2 (Active Comparator): Study group 2 will receive traditional treatment as the control group plus Kinesio tape on the popliteus muscle.
  Interventions: Other: Traditional Physical Therapy Treatment; Other: Kinesio Taping

INTERVENTIONS:
Other: Traditional Physical Therapy Treatment — Quadriceps strength, hip abduction strength, hip extension strength, hamstring stretch, gait training
Other: Popliteus Muscle Release — Myofascial release for the popliteus muscle
  Arms: Study Group 1
Other: Kinesio Taping — Kinesio tape on the popliteus muscle
  Arms: Study Group 2

SUMMARY:
The aim of the current study is to compare the effect of popliteus muscle release and Kinesio taping on pain intensity, function, dynamic balance, and quadriceps muscle strength in patients with patellofemoral pain syndrome.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome has been described as one of the most perplexing and clinically challenging chronic disorders.

Symptoms usually include diffuse pain originating from the anterior aspect of the patella and commonly along the medial aspect of the knee. It therefore limits daily activities that need loading on a flexed knee. There is a high incidence, especially among runners, with patellofemoral pain syndrome accounting for 46% of running-related injuries. However, the etiology of this disorder remains vague and controversial. This is reflected in the lack of consensus on how patellofemoral pain syndrome should be treated clinically. Patellofemoral pain syndrome participants have demonstrated abnormal gait patterns with decreased stance phase knee flexion, decreased walking velocity, and decreased muscle activity of the quadriceps musculature. Restoration of normal gait kinematics may be an important component of improving function.

The soft tissue manipulation decreased knee pain and improved muscle activity. Therefore, incorporating popliteus manipulation can be effective in the treatment of anterior knee pain.

Several systematic reviews and meta-analyses of Kinesio Taping treatment in different knee or musculoskeletal problems have been published in recent years. The support taping could reduce pain as an adjunct to traditional exercise therapy in patients with patellofemoral pain syndrome.

Kinesio Taping has a significant effect on pain reduction, motor function improvement, and muscle activity change.

So, the current study will help to determine the effect of myofascial release and Kinesio Taping of the popliteus muscle on patellofemoral pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders with an age range of 18-30 years old.
* minimum 3-month history of patellofemoral pain.
* a pain score for worst pain intensity during the previous week of 3 or more on a Visual Analog Scale (0-10, most pain).
* reproduced by at least two of the following activities: Stair ascent or descent, hopping, running, prolonged sitting, squatting, or kneeling and present on at least one of the following clinical tests: Compression of the patella or palpation of the patellar facets.

Exclusion Criteria:

* Clinical, x-ray, or MRI findings indicative of other specific pathology, including osteoarthritis, meniscal, ligament, or cartilage injury, or apophysitis.
* recurrent patellar subluxation or dislocation.
* cortisone use over an extended period of time.
* previous surgery to the knee joint; trauma to the knee joint affecting the presenting clinical condition.
* physiotherapy or other similar exercises for patellofemoral pain syndrome within the previous 3 months.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-01-10 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | It will be assessed at baseline and after 4 weeks.
  by visual analogue scale The visual analogue scale represents the pain range that a patient thinks they might experience. The line is typically 10 centimeters long, with anchor descriptors such as (in the pain context) "no pain" and "worst pain imaginable." The patient makes a mark reflecting his or her perception, and the distance from the left endpoint to the mark is measured in centimeters. Higher scores represent worse pain.
Knee Function | It will be assessed at baseline and after 4 weeks.
  by kujala scale The Arabic Kujala Patellofemoral Disorder scale, also called the anterior knee pain scale, is composed of 13 multiple-choice questions, each contributing to a total score ranging from 0 to 100. A higher score indicates better knee function and less pain, while a lower score reflects greater pain and disability.
Balance | It will be assessed at baseline and after 4 weeks.
  by Star Excursion Balance Test (SEBT)

SECONDARY OUTCOMES:
Quadriceps Strength | It will be assessed at baseline and after 4 weeks.
  by handheld dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Hafsa He Abdullah, MSc, Principal Investigator — Cairo University
Locations (1):
- Suez, Suez, Egypt

IPD SHARING:
Plan to Share IPD: No